CLINICAL TRIAL: NCT03367390
Title: An Early Feasibility Study to Evaluate the Functionality and Safety of an Automated Insulin Delivery System in Adult Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of an Automated Insulin Delivery System in Participants With Type 1 Diabetes Mellitus (T1DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16679; F3Z-MC-IOQS (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-12-05; First posted 2017-12-08 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AID System Containing Insulin Lispro (Experimental): The AID system is comprised of a continuous subcutaneous insulin infusion (CSII) pump component with a hybrid closed-loop control (HCLC) algorithm, and a continuous glucose monitor (CGM) component.
  Interventions: Device: AID System; Drug: Insulin Lispro

INTERVENTIONS:
Device: AID System — AID system
  Other Names: LY8888AU
Drug: Insulin Lispro — Individualized doses of insulin lispro administered via the AID system to maintain glycemic control, except during procedures designed to induce hyperglycemia and hypoglycemia.
  Other Names: LY275585

SUMMARY:
The Automated Insulin Delivery (AID) System is an investigational insulin delivery device being developed for use for participants with diabetes. The purpose of this study is to assess the safety of the AID system and to test whether the AID System functions as it was designed to.

This study will last approximately 12-18 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with T1DM for at least 2 years and who have used an insulin delivery system for at least 1 year
* Have a body mass index of 18.5 to 35 kilogram per meter squared
* Have a hemoglobin A1c level ≥6.0% and ≤9.0%

Exclusion Criteria:

* Have known allergies or history of hypersensitivity to insulin lispro
* Have had an episode of severe hypoglycemia within the past 6 months
* Have had more than 1 episode of diabetic ketoacidosis in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Show a Decrease or Suspension of Basal Insulin Delivery in Response to Hypoglycemia Challenges | Up to 4 hours post challenge
Number of Participants Who Show an Increase of Basal Insulin Delivery in Response to the Hyperglycemia Challenge | Up to 4 hours post challenge
Number of Participants Who Show a Resumption of Auto Mode Following Restored Continuous Glucose Monitoring (CGM) Connectivity | Up to 4 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Renton, Washington, United States

REFERENCES:
- See also: A Study of an Automated Insulin Delivery System in Participants With Type 1 Diabetes Mellitus (T1DM) — https://www.lillytrialguide.com/en-US/studies/type-1-diabetes/IOQS#?postal=